CLINICAL TRIAL: NCT06194916
Title: The Effect of Web-based Education Provided According to the Health Promotion Model on Self - Management in Epilepsy Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, ŞUHEDA ÜSTÜNDAĞ, science expert, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: AtaturkU-HMŞRLK-SU-01
Record Dates: First submitted 2023-12-22; First posted 2024-01-08 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2023-12

CONDITIONS: Epilepsy
Keywords: epilesy,education,self management
MeSH Terms: conditions — Epilepsy | interventions — Educational Status; Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- education group (Experimental): A 4-week web-based self-management training will be administered to epilepsy patients in the experimental group.
  Interventions: Other: Education
- Control Group (Active Comparator): routine interventions
  Interventions: Other: CONTROL GROUP

INTERVENTIONS:
Other: Education — A 4-WEEK SELF-MANAGEMENT TRAINING WILL BE PROVIDED THROUGH THE WEB-BASED TRAINING SITE.
  Arms: education group
Other: CONTROL GROUP — THEY WILL RECEIVE THE ROUTINE CARE GIVEN TO PATIENTS WITH EPILEPSY.
  Arms: Control Group

SUMMARY:
Epilepsy is a disease that requires long-term treatment and follow-up. Epilepsy To be successful in management, the educational needs of the patient must first be determined and the individual Treatment compliance should be increased by ensuring self-management of the disease.Interventions planned based on the model in patient education direct caregivers to specific goals and provide more planned, coordinated and safe care. The Health Promotion Model (HGM), developed by Nola Pender, is one of the models used to explain health protection and promotion behaviors. It is not aimed at preventing any disease or disability, but aims to improve health, in other words, to further increase the general health and well-being of the individual.

H0: Web-based education given to epilepsy patients according to the Health Promotion Model has no effect on self-management.

H1: Web-based education given to epilepsy patients according to the Health Promotion Model has an effect on self-management.

Research Inclusion Criteria:

1. Individuals who agree to participate in the research
2. Being over 18 years of age
3. Having been diagnosed with epilepsy for at least 1 year
4. Being able to use technological devices (phone, computer, tablet)
5. Having internet access,
6. Being able to speak Turkish,
7. Not having any additional disease
8. Being literate When starting the study, patients who apply to the outpatient clinic and meet the inclusion criteria will be given an explanation about the purpose of the research and how the research process will work. Then, written consent will be obtained indicating that they agree to participate in the study. Pretest data will be collected online. "Personal Information Form" and "Epilepsy Self-Management" scale will be used for individuals in the control and experimental groups to collect data.

In preparing the infrastructure of the web-based training program, a website called "Epilepsy Training Program" will be created with support from a professional computer engineering company. The training will include topics such as epilepsy, seizure management, medication management, safety management and lifestyle management. A training program consisting of presentations and videos will be offered on the website for a total of 4 weeks.

3 months after the training is completed, the "Epilepsy Self-Management Scale" will be applied to the experimental and control groups as a posttest.

DETAILED DESCRIPTION:
Epilepsy; It is a chronic neurological disease characterized by epileptic seizures that occur as a result of abnormal and excessive electrical discharge in cortical neurons, develop suddenly, are repetitive, and are not triggered by an identifiable event. Epilepsy is a disease that requires long-term treatment and follow-up. To be successful in the management of epilepsy, the educational needs of the patient must first be determined and the individual's compliance with the treatment must be increased by ensuring self-management of the disease.

Patient education is supporting the patient's independence to meet his or her own health needs. In a randomized controlled study, within the scope of a modular epilepsy education program, patients were given; Information was given about the etiology, epidemiology, diagnosis, treatment options, self-control, life with epilepsy and psychosocial dimensions of epilepsy, and it was determined that there was a significant increase in coping with the disease of the patients included in the program. In a randomized controlled study conducted in Iran, when looking at the effect of self-management training given to epilepsy patients with low education levels on medication compliance, it was found that medication compliance was significantly higher in the trained group.

Interventions planned based on the model in patient education direct caregivers to specific goals and provide more planned, coordinated and safe care. The Health Promotion Model (HGM), developed by Nola Pender, is one of the models used to explain health protection and promotion behaviors. It is not aimed at preventing any disease or disability, but aims to improve health, in other words, to further increase the general health and well-being of the individual. It has been reported that training based on SGM in various chronic diseases is effective in improving health behaviors. In a study examining the effect of patient education based on SGM on breast and cervical cancer early detection behaviors, it was reported that patients developed positive behavioral changes after the training. Again, in a study conducted to standardize diabetes education, an epilepsy management model was created based on SGM.

When starting the study, patients who apply to the outpatient clinic and meet the inclusion criteria will be given an explanation about the purpose of the research and how the research process will work. Then, written consent will be obtained indicating that they agree to participate in the study. Pretest data will be collected online. "Personal Information Form" and "Epilepsy Self-Management" scale will be used for individuals in the control and experimental groups to collect data.

In preparing the infrastructure of the web-based training program, a website called "Epilepsy Training Program" will be created with support from a professional computer engineering company. The training will include topics such as epilepsy, seizure management, medication management, safety management and lifestyle management. A training program consisting of presentations and videos will be offered on the website for a total of 4 weeks.

3 months after the training is completed, the "Epilepsy Self-Management Scale" will be applied to the experimental and control groups as a posttest.

Data Collection Tools:

Personal Information Form: It was created by the researcher as a result of literature review. It includes introductory sociodemographic characteristics of the patients and questions about the disease.

Epilepsy Self-Management Scale: Developed by Dilorio et al. (2004). A Turkish validity and reliability study was conducted by Yeni (2014). The scale consists of 38 items; It has five subscales that evaluate medication (10 items), safety (8 items), information (8 items), lifestyle (6 items) and seizure (6 items) management in individuals with epilepsy. It is evaluated in a 5-point Likert format and is scored between 1-5. 38 points is the minimum score that can be obtained from the scale, 190 points is the maximum score, and high scores indicate that individuals frequently use self-management behaviors. The Cronbach Alpha reliability coefficient of the Epilepsy Self-Management Scale was found to be 0.740.

Evaluation of Data: Data will be analyzed with SPSS for Windows 17 package program. Score average, percentages, standard deviation, and other analyzes deemed appropriate will be used when analyzing the data.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals who agree to participate in the research
2. Being over 18 years of age
3. Having been diagnosed with epilepsy for at least 1 year
4. Being able to use technological devices (phone, computer, tablet)
5. Having internet access,
6. Being able to speak Turkish,
7. Not having a psychiatric disease.

Exclusion Criteria:

* 1. Individuals who do not agree to participate in the research 2. Those under 18 years of age 3. Those with a psychiatric illness 4. Those who cannot use technological devices 5. Those who do not speak Turkish 6. Those diagnosed in less than 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Personal Information Form Epilepsy Self-Management Scale | pre-educationup to 4 weeks up to 8 weeks

SECONDARY OUTCOMES:
Epilepsy Self-Management Scale | 3 months after the education is completed

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code